CLINICAL TRIAL: NCT06744517
Title: Influence of Menstrual Cycle Phase on Metabolic and Performance Adaptations to Sprint Interval Training
Brief Title: Influence of Menstrual Cycle Phase on Adaptations to Sprint Interval Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Jenna Gillen, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HSREB50581
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: exercise; women
MeSH Terms: conditions — Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Follicular Phase Training (Active Comparator): Exercise training in the follicular phase (~days 1-14) of the participant's menstrual cycle
  Interventions: Other: Sprint Interval Training
- Luteal Phase Training (Experimental): Exercise training in the luteal phase (~days 15-28) of the participant's menstrual cycle
  Interventions: Other: Sprint Interval Training

INTERVENTIONS:
Other: Sprint Interval Training — 6 sessions of sprint interval training over 2 weeks. Each session involves 4-6 x 30 second Wingate sprints with 4 minutes of recovery in between on a stationary bike

SUMMARY:
Sprint interval training improves endurance performance and induces metabolic adaptations in muscle. Most research demonstrating these responses has been conducted in males, with limited studies evaluating changes to endurance performance and skeletal muscle oxidative capacity in females. Moreover, it is currently unknown if training in specific phases of the menstrual cycle influences adaptations to training. Thus, the purpose of the present study is to compare adaptations to 2 weeks of sprint interval training performed in the follicular vs. luteal phase of the menstrual cycle in healthy, eumenorrheic women.

DETAILED DESCRIPTION:
The primary purpose of the present study is to determine if menstrual cycle phase influences adaptations to 2 weeks of sprint interval training. Participants will be randomized to perform 6 sessions of sprint interval training over 2 weeks in either the Follicular Phase or Luteal Phase of their individual menstrual cycle. Blood and urine sampling will be used to confirm menstrual cycle phases. Training will involve 4-6 x 30-second Wingate sprints with 4 minutes of rest in between (~14-28 min per session). Before and after the training intervention, investigators will measure participant's aerobic and anaerobic performance, cardiorespiratory fitness and skeletal muscle outcomes. Performance and fitness measures are performed on on a stationary bike, and muscle outcomes are measured by taking a small amount of muscle from the vastus lateralis (thigh) muscle.

This study will advance knowledge on how the menstrual cycle influences adaptations to training in females

ELIGIBILITY:
Inclusion Criteria:

* Participating in 150 min of moderate-vigorous physical activity/week
* VO2peak of 'good' or above based on American College of Sport Medicine (ACSM) normative values(greater than 35.0ml/kg/min)
* Body mass index (BMI) between 18-27 kg/m2
* Performing 2-4 structured exercise sessions/week.
* Weight stable (within ± 2kg for at least 6 months)
* Non-smoker
* Menstrual cycle length of 27-35 days
* Minimal menstrual cycle length variability (less than 3 days)
* Ovulating monthly evidenced by a positive urinary luteinizing hormone surge
* Blood progesterone concentration greater than 16 nmol/L.

Exclusion Criteria:

* Hormonal contraceptive use within the last 3 months
* Polycystic ovarian syndrome (PCOS) or endometriosis
* Failure to meet MC verification criteria.
* Diagnosed with cardiovascular or metabolic disease, hyper- or hypogonadism, and/or PCOS
* The use of medication for managing blood glucose or lipid metabolism
* Current use of oral contraceptives or use within the last 3 months
* Irregular menstrual cycles (<27 days or >35 days)
* Pregnant or post-partum in the last 12 months, lactating or breast feeding within 3 months of the start of study, or menopausal
* Recreational smoking tobacco
* Inability to perform the study exercise protocols or follow the pre-trial dietary or physical activity controls
* Taking medications affecting substrate metabolism (corticosteroids or nSAIDs)
* Actively engaging in a low-carbohydrate diet (e.g., ketogenic, Atkins)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Endurance performance | Before and after 2 weeks of exercise training
  Time to completion and average power output during a 250kJ time trial

SECONDARY OUTCOMES:
Skeletal muscle mitochondrial content | Before and after 2 weeks of exercise training
  Measured via Western blotting
Skeletal muscle mitochondrial enzyme activity | Before and after 2 weeks of exercise training
  Measured via enzyme activity assays
Skeletal muscle capillarization | Before and after 2 weeks of exercise training
  Measured via immunofluorescence
Skeletal muscle lipid content | Before and after 2 weeks of exercise training
  Measured via immunofluorescence
Skeletal muscle protein synthesis | Before and after 2 weeks of exercise training
  Measured via the incorporation of a stable isotope tracer during the 2 weeks of training
Cardiorespiratory fitness | Before and after 2 weeks of exercise training
  Measured via a maximal exercise test on a cycle ergometer
Anaerobic exercise performance | Before and after 2 weeks of exercise training
  Power output during a Wingate anaerobic test

CONTACTS AND LOCATIONS:
Locations (1):
- Goldring Centre for High Performance Sport, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No